CLINICAL TRIAL: NCT02205229
Title: Compounded Pain Preparation Absorption Study (ComPPAS)
Brief Title: Compounded Pain Preparation Absorption Study
Acronym: ComPASS
Status: Suspended | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Medimix Specialty Pharmacy, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Medimix Pharm-03
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month

GROUPS / COHORTS (1):
- Patients receiving a topical compounded medication
  Interventions: Drug: Multi-ingredient, topical compounded medications

INTERVENTIONS:
Drug: Multi-ingredient, topical compounded medications

SUMMARY:
Single center, prospective, observational study to assess serum concentration of ingredients used in multi-ingredient, topical compounded medications from Medimix Specialty Pharmacy.

DETAILED DESCRIPTION:
Single center, prospective, observational, open-label, cohort study of participants that receive a combination topical pain medication from Medimix Specialty Pharmacy with no comparator group designed to assess serum concentration of ingredients used in multi-ingredient, topical compounded medications.

ELIGIBILITY:
Inclusion Criteria:

* Participants must apply and consistently use the supplied cream for 1 month at a prescribed
* Participants must be ≥ 30 and <65 years of age
* Participants must be able to provide sound written and verbal informed consent
* Participants must be diagnosed with an ICD9 code indicative of chronic pain

Exclusion Criteria:

* Participants must not have prior hypersensitivity or adverse events to any of the components in the customized prescription
* Participants must not be pregnant or breastfeeding
* Participants must not have used any study drug greater than 180 days from the day of Screening
* Participants must not be utilizing medications that may interact with those being used in the topical formulation as determined by the PI
* Participants must not be using any systemic medications that may influence drug serum concentrations of ingredients being used in the topical compound. These include medications from the same class of studied drugs or drugs that may falsely increase or decrease serum levels of the study drugs

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient between the ages of 30 and <65 years old not taking concomitant medications that may interact with study ingredients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of ingredients used in multi-ingredient, topical compounded medications | 1 Month

CONTACTS AND LOCATIONS:
Locations (1):
- Medimix Specialty Pharmacy, Jacksonville, Florida, United States